CLINICAL TRIAL: NCT06180018
Title: Modified TIP (Snodgrass) Using Interrupted Sutures in Hypospadias
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mahmoud mohamed kamel mohamed, director, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: modified TIP
Record Dates: First submitted 2023-11-09; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cases (Experimental): Using interrupted sutures
  Interventions: Other: interrupted sutures

INTERVENTIONS:
Other: interrupted sutures — Using interrupted sutures in repair of hypospadias by Snodgrass TIP repair

SUMMARY:
Using interrupted sutures in TIP technique by Snodgrass in repair of hypospadias instead of continuous sutures

ELIGIBILITY:
Inclusion Criteria:

* Midshaft , distal ,
* coronal hypospadias

Exclusion Criteria:

-

Ages: 6 Months to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Decreasing complications | 1 year
  New technique to decrease complications of this operation

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut, Asyut, Egypt